CLINICAL TRIAL: NCT03380468
Title: Adjuvant Chemotherapy Versus Observation in Fully Resected Stage I Lung Adenocarcinoma With High Risk of Post-operative Recurrence
Brief Title: Adjuvant Chemotherapy for High Risk Stage I Lung Adenocarcinoma
Acronym: ECTOP-1004
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Chief,department of thoracic surgery, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECTOP-1004
Record Dates: First submitted 2017-11-01; First posted 2017-12-21 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Lung Neoplasms
Keywords: Lung adenocarcinoma; adjuvant chemotherapy
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma of Lung | interventions — Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cisplatin plus pemetrexed (Experimental): Drug: cisplatin 75mg/m2 iv Drug: pemetrexed 500mg/m2 iv
  Interventions: Drug: cisplatin plus pemetrexed
- Observation (No Intervention): Observation and follow up only

INTERVENTIONS:
Drug: cisplatin plus pemetrexed — cisplatin 75mg/m2 iv; pemetrexed 500mg/m2 iv
  Arms: Cisplatin plus pemetrexed

SUMMARY:
This is a clinical trial from Eastern Cooperative Thoracic Oncology Project (ECTOP), numbered as ECTOP-1004. Solid subtype, micropapillary subtype, vascular involvement, pleural involvement and low differentiation are high risk factors of post-operative recurrence for early-stage lung adenocarcinoma patients. The purpose of this clinical trial is to determine whether the widely used adjuvant chemotherapy strategy cisplatin/ pemetrexed is more effective than no further treatment for Stage pI lung adenocarcinoma patients with high post-operative recurrence risk - in terms of no dose related toxicities, premature treatment withdrawal or death.

DETAILED DESCRIPTION:
Background:

Management of lung cancer varies according to the clinical and pathological stage. For stage I lung adenocarcinoma, radical surgery is the preferred initial treatment and adjuvant chemotherapy is usually not recommended due to a fine prognosis and relatively low post-operative recurrence rate. Still, a number of stage pI patients will suffer a relapse after surgery, among which are highly associated with solid subtype, micropapillary subtype, vascular involvement, pleural involvement and low differentiation. Recently, some retrospective researches have shown a significant survival benefit of adjuvant chemotherapy for such stage pI high-recurrent-risk patients, but there lacks evidence from prospective randomized clinical trails.

Objective:

1. Major: to compare disease free survival and over all survival of fully resected stage pI high-recurrent-risk patients from both arms (adjuvant chemotherapy vs. observation)
2. To assess the safety and efficacy of chemotherapy regimen cisplatin plus pemetrexed to fully resected stage pI high-recurrent-risk patients.
3. To collect clinical pathological characteristics and prognosis information of stage pI patients with solid subtype, micropapillary subtype, vascular involvement, pleural involvement and low differentiation.
4. To determine the association among age, gender, smoking history, pathological subtypes, histological differentiation, pleural involvement, vascular involvement and driving mutations.

Randomization:

Each of the patients enrolled will be recorded in the computer system. Blank randomization will be done using a digital randomization software, at least 1 week before the first time of chemotherapy or observation.

Prechemotherapy assessment: For all the patients enrolled, the postoperative physical or laboratory examination should be equally qualified no matter which group they will be in. For Group Adjuvant Chemotherapy patients, they will receive laboratory examinations before chemotherapy to test blood cells and liver function in consideration of safety as routine.

Follow up:

Patients will be followed up per 4 months for the first three years and each six months for the forth to fifth years during the research. Lung multi-detector row computed tomography (MDCT) and abdominal ultrasonography tests will be done twice a year; bone SPECT scan and enhanced brain MRI scan will be conducted per year routinely. Patients will be suggested to continue the annual follow-up after the research.

Main research variables:

Primary end point: Disease free survival in the two arms

Secondary endpoints:

1. Overall survival
2. Recurrence pattern: Locoregional recurrence, metastatic recurrence, or both
3. Quality of life: assessed with Eastern Cooperative Oncology Group- quality of life questionnaire(EORTC QLQ-C30/- LC13) scale.

This study is recognized in our institute as "Eastern Cooperative Thoracic Oncology Projects (ECTOP-1004)"

ELIGIBILITY:
Inclusion Criteria:

1. Stage pI lung adenocarcinoma confirmed through formalin-fixed paraffin-embedded tumor tissue, complete resection with mediastinal lymph node dissection
2. Meet one of following conditions: a, Solid predominant adenocarcinomas; b, micropapillary predominant adenocarcinoma; c, low differentiation, unable to identify histological subtypes; d, pleural involvement; e, vascular involvement with solid subtype component or micropapillary component.
3. Aged 18-70 years old.
4. Eastern Cooperative Oncology Group score standard (ECOG) status 0-1.
5. Medical condition permits adjuvant chemotherapy.
6. Patients accept the clinical trial protocol and Informed Consent Form (ICF) signed.

Exclusion Criteria:

1. Concurrent other malignancies
2. Prior chemotherapy and/or radiation therapy for lung cancer
3. Central type lung cancer
4. Concurrent other unresected suspicious nodules or masses in lung
5. Medical condition that will not permit treatment or follow up according to the protocol, or ECOG status >1.
6. Pregnant or nursing women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival (RFS) | up to 5 years
  from date of randomization until the date of showing signs of relapse, including evidence of medical image or pathology.

SECONDARY OUTCOMES:
Overall survival (OS) | up to 5 years
  from date of randomization until the date of death from any cause, withdrawal of consent, or the end of the study.

OTHER OUTCOMES:
Recurrence pattern | up to 5 years
  locoregional recurrence, metastatic recurrence, or both.
Quality of life | up to 5 years
  assessed with Eastern Cooperative Oncology Group-quality of life questionnaire(EORTC QLQ-C30/- LC13) scale.
  Discription of EORTC QLQ-C30/- LC13:
  The full name of the scale is Eastern Cooperative Oncology Group- quality of life questionnaire, including a core scale (EORTC QLQ-C30, version 3.0) and a module specified for lung cancer (EORTC QLQ- LC13). The scale is authorized by Quality of Life Department, EORTC Headquarters (Avenue E Mounier 83 - B11, 1200 Brussels BELGIUM) for scientific research.
  The scale ranges in score from 0 to 100. A higher score represents a a better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Haiquan Chen, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Kelsey CR, Marks LB, Hollis D, Hubbs JL, Ready NE, D'Amico TA, Boyd JA. Local recurrence after surgery for early stage lung cancer: an 11-year experience with 975 patients. Cancer. 2009 Nov 15;115(22):5218-27. doi: 10.1002/cncr.24625. PMID 19672942
- [Background] Zhang Y, Li J, Wang R, Li Y, Pan Y, Cai D, Hu H, Li H, Ye T, Luo X, Zhang Y, Li B, Shen L, Sun Y, Chen H. The prognostic and predictive value of solid subtype in invasive lung adenocarcinoma. Sci Rep. 2014 Nov 24;4:7163. doi: 10.1038/srep07163. PMID 25418354
- [Background] Zhang Y, Wang R, Cai D, Li Y, Pan Y, Hu H, Wang L, Li H, Ye T, Luo X, Zhang Y, Li B, Shen L, Sun Y, Chen H. A comprehensive investigation of molecular features and prognosis of lung adenocarcinoma with micropapillary component. J Thorac Oncol. 2014 Dec;9(12):1772-8. doi: 10.1097/JTO.0000000000000341. PMID 25226429
- [Background] Yoshizawa A, Motoi N, Riely GJ, Sima CS, Gerald WL, Kris MG, Park BJ, Rusch VW, Travis WD. Impact of proposed IASLC/ATS/ERS classification of lung adenocarcinoma: prognostic subgroups and implications for further revision of staging based on analysis of 514 stage I cases. Mod Pathol. 2011 May;24(5):653-64. doi: 10.1038/modpathol.2010.232. Epub 2011 Jan 21. PMID 21252858
- [Background] Shimada Y, Saji H, Yoshida K, Kakihana M, Honda H, Nomura M, Usuda J, Kajiwara N, Ohira T, Ikeda N. Pathological vascular invasion and tumor differentiation predict cancer recurrence in stage IA non-small-cell lung cancer after complete surgical resection. J Thorac Oncol. 2012 Aug;7(8):1263-70. doi: 10.1097/JTO.0b013e31825cca6e. PMID 22673056
- [Background] Al-Alao BS, Gately K, Nicholson S, McGovern E, Young VK, O'Byrne KJ. Prognostic impact of vascular and lymphovascular invasion in early lung cancer. Asian Cardiovasc Thorac Ann. 2014 Jan;22(1):55-64. doi: 10.1177/0218492313478431. Epub 2013 Sep 4. PMID 24585645
- [Background] Chen YY, Huang TW, Tsai WC, Lin LF, Cheng JB, Lee SC, Chang H. Lymphovascular space invasion and tumor differentiation are predictors for postoperative recurrence in patients with pathological stage I nonsmall cell lung cancer. J Chin Med Assoc. 2014 Aug;77(8):416-21. doi: 10.1016/j.jcma.2014.05.008. Epub 2014 Jul 12. PMID 25028298
- [Background] Park C, Lee IJ, Jang SH, Lee JW. Factors affecting tumor recurrence after curative surgery for NSCLC: impacts of lymphovascular invasion on early tumor recurrence. J Thorac Dis. 2014 Oct;6(10):1420-8. doi: 10.3978/j.issn.2072-1439.2014.09.31. PMID 25364519
- [Background] Yano M, Sasaki H, Moriyama S, Kawano O, Hikosaka Y, Fujii Y. Prognostic factors of pathologic stage IB non-small cell lung cancer. Ann Thorac Cardiovasc Surg. 2011;17(1):58-62. doi: 10.5761/atcs.cr.09.01481. PMID 21587131
- [Background] Huang H, Wang T, Hu B, Pan C. Visceral pleural invasion remains a size-independent prognostic factor in stage I non-small cell lung cancer. Ann Thorac Surg. 2015 Apr;99(4):1130-9. doi: 10.1016/j.athoracsur.2014.11.052. Epub 2015 Feb 20. PMID 25704861
- [Background] Jiang L, Liang W, Shen J, Chen X, Shi X, He J, Yang C, He J. The impact of visceral pleural invasion in node-negative non-small cell lung cancer: a systematic review and meta-analysis. Chest. 2015 Oct;148(4):903-911. doi: 10.1378/chest.14-2765. PMID 25675151
- [Background] Butts CA, Ding K, Seymour L, Twumasi-Ankrah P, Graham B, Gandara D, Johnson DH, Kesler KA, Green M, Vincent M, Cormier Y, Goss G, Findlay B, Johnston M, Tsao MS, Shepherd FA. Randomized phase III trial of vinorelbine plus cisplatin compared with observation in completely resected stage IB and II non-small-cell lung cancer: updated survival analysis of JBR-10. J Clin Oncol. 2010 Jan 1;28(1):29-34. doi: 10.1200/JCO.2009.24.0333. Epub 2009 Nov 23. PMID 19933915
- [Background] Strauss GM, Herndon JE 2nd, Maddaus MA, Johnstone DW, Johnson EA, Harpole DH, Gillenwater HH, Watson DM, Sugarbaker DJ, Schilsky RL, Vokes EE, Green MR. Adjuvant paclitaxel plus carboplatin compared with observation in stage IB non-small-cell lung cancer: CALGB 9633 with the Cancer and Leukemia Group B, Radiation Therapy Oncology Group, and North Central Cancer Treatment Group Study Groups. J Clin Oncol. 2008 Nov 1;26(31):5043-51. doi: 10.1200/JCO.2008.16.4855. Epub 2008 Sep 22. PMID 18809614
- [Background] Luo J, Huang Q, Wang R, Han B, Zhang J, Zhao H, Fang W, Luo Q, Yang J, Yang Y, Zhu L, Chen T, Cheng X, Wang Y, Zheng J, Wu H, Xia W, Chen H. Prognostic and predictive value of the novel classification of lung adenocarcinoma in patients with stage IB. J Cancer Res Clin Oncol. 2016 Sep;142(9):2031-40. doi: 10.1007/s00432-016-2192-6. Epub 2016 Jul 5. PMID 27379889
- [Background] Tsao MS, Marguet S, Le Teuff G, Lantuejoul S, Shepherd FA, Seymour L, Kratzke R, Graziano SL, Popper HH, Rosell R, Douillard JY, Le-Chevalier T, Pignon JP, Soria JC, Brambilla EM. Subtype Classification of Lung Adenocarcinoma Predicts Benefit From Adjuvant Chemotherapy in Patients Undergoing Complete Resection. J Clin Oncol. 2015 Oct 20;33(30):3439-46. doi: 10.1200/JCO.2014.58.8335. Epub 2015 Apr 27. PMID 25918286
- [Background] Liu CH, Peng YJ, Wang HH, Chen YC, Tsai CL, Chian CF, Huang TW. Heterogeneous prognosis and adjuvant chemotherapy in pathological stage I non-small cell lung cancer patients. Thorac Cancer. 2015 Sep;6(5):620-8. doi: 10.1111/1759-7714.12233. Epub 2015 Feb 27. PMID 26445611
- [Background] Park SY, Lee JG, Kim J, Byun GE, Bae MK, Lee CY, Kim DJ, Chung KY. Efficacy of platinum-based adjuvant chemotherapy in T2aN0 stage IB non-small cell lung cancer. J Cardiothorac Surg. 2013 Jun 11;8:151. doi: 10.1186/1749-8090-8-151. PMID 23759129
- [Background] Tsuchiya T, Akamine S, Muraoka M, Kamohara R, Tsuji K, Urabe S, Honda S, Yamasaki N. Stage IA non-small cell lung cancer: vessel invasion is a poor prognostic factor and a new target of adjuvant chemotherapy. Lung Cancer. 2007 Jun;56(3):341-8. doi: 10.1016/j.lungcan.2007.01.019. Epub 2007 Mar 9. PMID 17350137
- [Background] Zhang H, Lu C, Lu Y, Yu B, Lv F, Zhu Z. The predictive and prognostic values of factors associated with visceral pleural involvement in resected lung adenocarcinomas. Onco Targets Ther. 2016 Apr 20;9:2337-48. doi: 10.2147/OTT.S100965. eCollection 2016. PMID 27143929
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390